CLINICAL TRIAL: NCT03875664
Title: Extended Release Local Anesthetic for Postsurgical Pain After Posterior Colporrhaphy and Perineorrhaphy: A Randomized Controlled Study
Brief Title: Extended Release Local Anesthetic for Postsurgical Pain After Posterior Colporrhaphy and Perineorrhaphy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00024327
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Results first posted 2020-05-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2020-05

CONDITIONS: Postoperative Pain
Keywords: liposomal bupivacaine; posterior repair
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Receives 20 mL liposomal bupivacaine expanded with 10 mL of injectable sterile normal saline solution (0.9%) for a total of 30 mL injected in the posterior vaginal compartment in a standardized technique
  Interventions: Drug: Liposomal bupivacaine
- Placebo (Placebo Comparator): Receives 30 mL of injectable sterile normal 0.9% saline solution injected in the posterior vaginal compartment in a standardized technique
  Interventions: Drug: Placebo - injection

INTERVENTIONS:
Drug: Liposomal bupivacaine — Extended-release local anesthetic
  Other Names: EXPAREL 266 mg
  Arms: Intervention
Drug: Placebo - injection — Injectable normal saline solution
  Arms: Placebo

SUMMARY:
The specific aim of this randomized double-blind clinical trial is to evaluate the effect of intraoperative infiltration of liposomal bupivacaine at the time of posterior colporrhaphy and/or perineorrhaphy on postsurgical pain scores during the first 72 hours after surgery as measured by visual analog scales (VAS) for patients undergoing surgery for pelvic organ prolapse. Study subjects are randomized to 30 mL of liposomal bupivacaine versus 30 mL of injectable normal saline administered in a standardized technique into the posterior vaginal compartment at the time of posterior repair and/or perineorrhaphy.

DETAILED DESCRIPTION:
Liposomal bupivacaine (EXPAREL; Pacira Pharmaceuticals, San Diego, CA) is an extended release local anesthetic approved by the Food and Drug Administration since 2011 for the treatment of postsurgical pain. It is a multivesicular liposomal delivery system, consisting of a liquid bupivacaine core encapsulated by a phospholipid shell. This delivery technology allows for the slow, sustained release of bupivacaine over at least 72 hours.

Liposomal bupivacaine has been studied extensively in the general surgery and orthopedic surgery literature. Specifically, infiltration of liposomal bupivacaine after excisional hemorrhoidectomy has been shown to significantly lower postsurgical pain scores, decrease total postoperative opioid requirements, increase the number of patients who do not require any opioids after surgery, meaningfully delay the median time to first opioid use, and improve patient satisfaction with overall perioperative analgesia.

Posterior colporrhaphy and perineorrhaphy are pelvic reconstructive surgical procedures that are associated with significant postsurgical localized pain resulting from surgical incisions. Investigators hypothesize this localized postsurgical pain will benefit from treatment with an extended release local anesthetic formulation similar to hemorrhoidectomy. Intraoperative infiltration of a standard local anesthetic during posterior repair and perineorrhaphy has been shown to improve early analgesia and facilitate early postoperative recovery. These findings reiterate the need for studies investigating a slow-release, longer-acting local anesthetic formulation for patients undergoing posterior repair and/or perineorrhaphy - one that ideally can be integrated into an evidence-based, opioid-sparing postsurgical pain management regimen to improve perioperative care for the steadily growing pelvic reconstructive surgical patient population.

The primary study objective is to evaluate the effect of intraoperative infiltration of liposomal bupivacaine at the time of posterior colporrhaphy and/or perineorrhaphy on postsurgical pain scores during the first 72 hours after surgery as measured by visual analog scales (VAS).

Secondary objectives include to evaluate total opioid consumption during the first 72 postoperative hours, to evaluate patient satisfaction with postoperative analgesia, to evaluate time to first opioid administration postoperatively, to evaluate hospital length of stay, to evaluate length of stay in post-anesthesia care unit (PACU), to evaluate total hospital costs, to evaluate time to first bowel movement postoperatively, to evaluate rate of postoperative nausea and vomiting, to evaluate time to successful voiding trial, and to evaluate proportion of patients discharged home with a Foley catheter.

Patients will be approached for participation preoperatively and randomized in the operating room to either liposomal bupivacaine or injectable normal saline administered into the posterior vaginal compartment in a standardized technique. All concurrent minimally invasive pelvic reconstructive surgical procedures are allowed. Randomization will be stratified for abdominal versus purely vaginal surgery. Perioperative care is standardized. Data will be abstracted from the medical record. Additionally, subjects will be discharged home with a medication diary and pain scales. Subjects will record their pain every morning and every evening for the first 72 hours after surgery. Subjects will complete a satisfaction survey at their 2 week postoperative visit. Adverse postoperative outcomes will be collected for 30 days after surgery.

The study is powered to detect a 20 mm difference in a 100 mm visual analog scale for pain.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking women ages 18 and older undergoing posterior repair and/or perineorrhaphy at our institution for pelvic organ prolapse

Exclusion Criteria:

* Planned regional anesthesia
* Allergy or contraindication to bupivacaine
* Allergy or contraindication to opioids
* Allergy or contraindication to non-steroidal medications
* Planned laparotomy
* Chronic pain diagnosis and/or chronic narcotic use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study involves women undergoing surgery for pelvic organ prolapse
Enrollment: 72 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Evans, MD, Principal Investigator — Women's Center for Pelvic Health
Locations (1):
- Women's Center for Pelvic Health, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excluded after enrollment if intraoperative decision made not to perform posterior colporrhaphy or perineorrhaphy.
Period: Overall Study
Arm/Group | Intervention | Placebo
Started | 37 | 35
Completed | 37 (vaginal surgery n=18; vaginal + abdominal surgery n=19) | 35 (Vaginal surgery n=18; vaginal + abdominal surgery n=17)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Placebo | Total
Number analyzed (Participants) | 37 | 35 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (13.5) | 61 (26.7) | 62.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 35 | 72
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 36 | 35 | 71
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 34 | 35 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain
Description: As measured by a 100 mm Visual Analog Scale (VAS). This scale ranges from 0-100 mm with 0 mm indicating no pain and 100 mm indicating the most pain. The study is powered to detect a decrease in postoperative pain by 20 mm on this scale, which is considered to be a clinically meaningful difference in prior studies. Results will be reported as mean pain scores at each time point (night of surgery, morning and evening for the first 72 hours after surgery, i.e. until postoperative day#3).
Time Frame: Night of surgery (POD#0), POD#1 morning, POD#1 evening, POD#2 morning, POD#2 evening, POD#3 morning, POD#3 evening
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 37 | 35
mm
  POD#0 evening | 1.9 [0 to 2.4] | 1.3 [0 to 4.3]
  POD#1 morning | 2.0 [0 to 4.1] | 1.9 [0 to 3.4]
  POD#1 evening | 2.9 [0 to 4.9] | 2.5 [0 to 3.5]
  POD#2 morning | 3.1 [0 to 6.5] | 2.4 [0 to 4.6]
  POD#2 evening | 2.3 [0 to 6.6] | 1.9 [0 to 4.2]
  POD#3 morning | 1.7 [0 to 3.5] | 1.9 [0 to 3.4]
  POD#3 evening | 2.3 [0 to 4.9] | 1.6 [0 to 4.6]

2. Secondary Outcome: Number of Participants Reporting Satisfaction With Pain Control
Description: As measured by a 5-question satisfaction survey administered at a 2 week postoperative visit. The survey includes Likert scale responses ranging from very unsatisfied to very satisfied with the surgical experience and specifically analgesia. "Patient Satisfaction" was defined as response "satisfied" or "very satisfied" on the Likert Scale. Average responses will be reported.
Time Frame: 2 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 37 | 35
Participants | 32 | 33

3. Secondary Outcome: Time to First Opioid Administration
Description: Median time until first opioid administered after surgery
Time Frame: Assessed up to 72 hours after surgery
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 37 | 35
minutes | 89.5 [60 to 219] | 68 [60 to 234]

4. Secondary Outcome: Total Opioid Administration
Description: Measured in milligram morphine equivalents
Time Frame: Cumulatively, over a time period of 72 hours after surgery
Measure: Mean (Standard Deviation); unit: mme
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 37 | 35
mme | 37.5 (40) | 37.5 (43.5)

5. Secondary Outcome: Number of Antiemetic Doses Required Per Participant While Inpatient
Description: Number of as-needed antiemetic doses patient received while in the hospital after surgery
Time Frame: Cumulatively, over a time period of 72 hours after surgery
Measure: Median (Inter-Quartile Range); unit: doses
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 37 | 35
doses | 2 [1 to 2] | 3 [1 to 3]

6. Secondary Outcome: Hospital Length of Stay
Description: Total length of hospital stay measured in hours, including readmissions
Time Frame: Assessed until 30 days after surgery
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 37 | 35
hours | 21.9 (20) | 24 (19.6)

7. Secondary Outcome: Length of Stay in Post-anesthesia Care Unit (PACU)
Description: Total length of stay in PACU measured in minutes
Time Frame: Assessed up to 72 hours after surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 37 | 35
minutes | 100 (61) | 93 (40)

8. Secondary Outcome: Number of Participants Who Had a Bowel Movement Within the First 3 Postoperative Days
Description: As recorded by patient - patients were asked each postoperative day (i.e. POD#0, POD#1, POD#2, POD#3) if they had a bowel movement that day, yes or no.
Time Frame: 72 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 37 | 35
Participants | 22 | 23

9. Secondary Outcome: Voiding Trial Failures
Description: Proportion of patients discharged home with Foley catheters after failed voiding trials in the hospital
Time Frame: 2 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 37 | 35
Participants | 15 | 19

10. Secondary Outcome: Number of Patients With Adverse Events
Description: Total adverse postoperative events
Time Frame: Assessed until 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 37 | 35
Participants | 6 | 11
Statistical Analysis 1: Comparison: Intervention vs Placebo; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 30 days
Description: We also investigated postoperative complications defined by the American College of Surgeon's National Surgical Quality Improvement Program (NSQIP).
  Adverse events were collected by chart review within 30 days of surgery. Charts were independently reviewed by 2 study personal for accuracy.
Arm/Group | Intervention | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/35
Other Adverse Events (participants affected / at risk) | 6/37 | 11/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=37) | Placebo (N=37)
Urinary Tract Infections (Infections and infestations) | 4 (4) | 9 (9) — 9 urinary tract infections in placebo group; 4 urinary tract infections in liposomal bupivacaine group
Hospital readmission (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Return to operating room (Surgical and medical procedures) | 0 (0) | 1 (1) — For midurethral sling revision

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT03875664/Prot_SAP_001.pdf
  • Informed Consent Form (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT03875664/ICF_002.pdf